CLINICAL TRIAL: NCT02801838
Title: Feasibility and Validity of an Observational Scale as a Surrogate of Dyspnea in Non-communicating Patients in the Intensive Care Unit (ICU): DYS-NOC
Brief Title: Validation of an Observational Scale of Dyspnea in Non-communicating Patients in the ICU
Acronym: DYS-NOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association pour le Développement et l'Organisation de la Recherche en Pneumologie et sur le Sommeil (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ADOREPS_2
Record Dates: First submitted 2016-05-06; First posted 2016-06-16 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Dyspnea
Keywords: Inspiratory muscles; Patient-ventilator interaction; Electromyogram; Mechanical ventilation
MeSH Terms: conditions — Dyspnea | interventions — Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ventilator settings, morphine titration (Experimental): First, ventilator settings optimization and when the clinician judges necessary (remains discomfortable), opioid titration with a maximum of 10mg of morphine
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Morphine — If the physician in charge of the patients judges it necessary, after the optimization of the ventilators settings, if the patient remains uncomfortable, a second therapeutic intervention using a maximum of 10mg morphine titration may be performed. After this second therapeutic intervention, a third non-verbal measure of respiratory discomfort will be performed with the IC-RDOS. Concomitantly, EEG and EMG will be again recorded over a of 15-minutes period.
  Other Names: Morphine sulfate

SUMMARY:
Background : Dyspnea is common and severely impact mechanically ventilated patients outcomes in intensive care unit (ICU). Recognize, measure and treat dyspnea have become current major therapeutic challenge. Its measurement involves a self-assessment by the patient, and by definition, a certain level of communication. Consequently, a large proportion of the ICU-population (non-communicating) misses its evaluation and potential benefits associated with its control. In other hand, electrophysiological markers that help to detect and quantify dyspnea regardless of the patient's cooperation, has been developed and validated as dyspnea surrogate, namely: 1) the electromyographic (EMG) activity of extra diaphragmatic inspiratory muscles and 2) the premotor inspiratory potentials (PIP) detected on the electroencephalogram (EEG). Because of its complex implementation in daily practice the research team has developed alternatively a behavioral score called IC-RDOS that provides reliable dyspnea assessment also without patient participation. Validated in conscious patients, it has not been yet validated in non-communicating patients.

Hypothesis : The IC-RDOS is valid for non-communicating ventilated patients and allows a simple and reliable assessment of dyspnea in this specific population.

Objective : To validate the IC-RDOS in non-communicating ICU patients under mechanical ventilation, using comparison with the tools validated for reliable measure of dyspnea in non-communicating patients (EMG, EEG).

Patients and Methods: In 40 patients will be collected simultaneously IC-RDOS, PIP (EEG) and electromyographic activity of three extra diaphragmatic inspiratory muscles (scalene, parasternal and Alae nasi) before and after intervention therapy aiming at reduce dyspnea (ventilator settings or pharmacological intervention), initiated by the clinician in charge of the patient.

Expected results : Observe a strong positive correlation between the IC-RDOS and electrophysiological markers (amplitude of the electromyogram and presence and magnitude of PIP). Observe a correlation between changes in the IC-RDOS and the electrophysiological markers after therapeutic interventions.

Optimizing patient comfort is a prominent concern in the ICU. By optimizing the detection and quantification of dyspnea in non-communicating patients, this study should ultimately improve the management and "the better living" of ventilated patients in intensive care

DETAILED DESCRIPTION:
INTRODUCTION

It becomes clear that dyspnea is becoming a major matter of concern in ICU mechanically ventilated patients. As this is the case for pain, addressing dyspnea in ICU patients therefore appears highly clinically relevant. This requires focused awareness from caregivers and patient cooperation. Indeed, because dyspnea involves the sensory identification of afferent signals by the brain and their cognitive and affective processing, its characterization depends on self-report. Clinical signs of "respiratory distress" and self-perceived dyspnea can be disconnected, setting a limitation to identifying dyspnea in many ICU patients whose ability to communicate verbally is impaired. Nevertheless, a link does exist between dyspnea and certain observable signs. A respiratory distress observation scale (RDOS) has been validated as a surrogate for self-reported dyspnea in the palliative care setting.

In ICU patients, the research team has recently developed and validated a 5-items intensive care (IC)-RDOS (heart rate, neck muscles use during inspiration, abdominal paradox, fear expression, supplemental oxygen). The findings validate IC-RDOS as potential surrogates of dyspnea in the ICU, proving the concept that observation scales can be useful in this context. Indeed, IC-RDOS had a high sensitivity and specificity to predict a dyspnea-VAS ≥4. However, IC-RDOS is only validated in aware patients and its clinical usefulness in "non communicating" patients still need to be demonstrated.

Addressing dyspnea in "non-communicating" patients is challenging since these patients cannot self-report dyspnea. However, it does not mean at all that they do not experience dyspnea. Indeed, "non-communicating" and "communicating" mechanically ventilated patients are equally submitted to risk factors for dyspnea. Moreover, ignoring dyspnea in a "non-communicating" patient may increase the risk of inadequate ventilator settings, which could in turn even increase dyspnea.

To address this issue, the research team and others have developed and validated reliable electrophysiological makers that help to detect and quantify dyspnea regardless of the patient's self-report ability: 1) the electromyographic (EMG) activity of extra diaphragmatic inspiratory muscles and 2) the premotor inspiratory potentials (PIP) detected on the electroencephalogram (EEG).

1. The EMG activity of three extra diaphragmatic inspiratory muscles (scalene, parasternal intercostal muscles and Alae nasi) is a reliable surrogate of the load capacity balance in healthy subjects and in patients with a respiratory disease. In ICU patients, this EMG activity is significantly correlated with the dyspnea-VAS.
2. The application of an inspiratory resistive load to healthy subjects results in the activation of the pre-motor cortex detected by EEG recording named pre-inspiratory potential (PIP).

OBJECTIVE

The objective of the study is to validate the IC-RDOS as a surrogate of dyspnea in "non-communicating" mechanically ventilated patients in the ICU. To achieve this goal, the IC-RDOS will be compared to two electrophysiological tools that are validated for the assessment of dyspnea in "non-communicating" patients, the EMG of extra diaphragmatic inspiratory muscles and the PIP on the EEG. This comparison will be performed before and after a therapeutic intervention aiming at reduces dyspnea because the concomitant variation of the scale and of the neurophysiological markers is required to validate the reliability of the scale.

The specific aims will be to simultaneously collect the IC-RDOS, PIP and the EMG activity of the Scalene, Parasternal intercostal muscles and Alae nasi,

1. Before any intervention,
2. And after an intervention aiming at reduce dyspnea.

STUDY DESIGN

A first non-verbal measure of respiratory discomfort will be achieved through the IC-RDOS by the experimenter. Concomitantly, EEG and EMG will be recorded over a 15-minutes period.

The therapeutic interventions aiming at reduce dyspnea will be performed by the clinician in charge of the patient, who will be strictly independent of the experimenter. This intervention could be a change in ventilator settings or an administration of a pharmacological agent. The nature of the intervention will be recorded but will remain blinded to the experimenter.

After the therapeutic intervention, a second non-verbal measure of respiratory discomfort will be performed with the IC-RDOS. Concomitantly, EEG and EMG will be recorded over a 15-minutes period.

If the physician in charge of the patients judges it necessary, a second therapeutic intervention may be performed. After this second therapeutic intervention, a third non-verbal measure of respiratory discomfort will be performed with the IC-RDOS. Concomitantly, EEG and EMG will be again recorded over a of 15-minutes period.

EXPECTED RESULTS

Observe a strong positive correlation between non-verbal numerical evaluation of dyspnea by the IC-RDOS and the amplitude of the EMG activity of the three extra diaphragmatic inspiratory muscles.

Observe a significant positive association between the presence and the amplitude of a PIP and the value of the IC-RDOS.

Observe a significant association between the change in the IC-RDOS and the respective changes in the EMG activity of extra diaphragmatic inspiratory muscles and in the amplitude of the PIP.

Observe a decrease in the proportion of dyspneic patients after therapeutic intervention. Observe an average relative reduction of the IC-RDOS after therapeutic intervention.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included as soon as all the following criteria will be met.

* Invasive mechanical ventilation for > 24 h.
* All cycles triggered by the patient.
* "Non-communicating" patient, defined as a score < -1 on the Richmond Agitation and Sedation Scale (RASS) [1].
* Suspicion by the clinician in charge of the patient of a dyspnea by at least two of the four following elements: tachypnea > 25 cycles/min ; suprasternal or supraclavicular draw ; abdominal paradox on inspiration ; facial discomfort expression (facial rating scale).
* Decision by the physician in charge of the patient to make an intervention in order to reduce dyspnea. This intervention will consist either in change in ventilator settings or in the administration of pharmacologic agents that reduce dyspnea, such as opioids.

Exclusion Criteria:

Exclusion criteria will be as follows.

* Age < 18 years.
* Pregnancy.
* Severe acquired or congenital neuropathy or myopathy that could affect the physical or behavioural manifestations of dyspnea and the collection of EMG activity of inspiratory extra diaphragmatic muscles.
* Central neurological disease that may alter the collection of PIP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-02-23 (Actual); Primary Completion 2017-02-23 (Actual); Study Completion 2017-07-28 (Actual)

PRIMARY OUTCOMES:
Respiratory comfort with IC-RDOS | in real time, during the procedure
  Quantification of dyspnea:
  Dyspnea will be quantified with the ICU Respiratory distress operating scale.

SECONDARY OUTCOMES:
EMG signals of extradiaphragmatic muscles | in real time, during the procedure
  EMG signals will be collected using surface electrodes (Kendall, Tyco Healthcare, Germany).
  Bilateral para-sternal intercostal-target recordings will be obtained from the second intercostal space, close to the sternum. Bilateral scalene-targeted recordings will be obtained in the posterior triangle of the neck at the level of the cricoid cartilage. Alae nasi-targeted recordings will be obtained by placing one electrode on each nostril.
  A distance of 2 cm separates the electrode pairs. The impedance must remain below 2000 Ω. Cables connected to the electrodes will be fixed with adhesive tape to prevent the occurrence of artifacts related to the movement of the upper limbs. All these signals will be recorded at a sampling frequency of 1000 Hz (PowerLab, AD Instruments, Castle Hill, Australia).
Airways flow | in real time, during the procedure
  Airways flow will be measured with a pneumotachograph
Airways pressure | in real time, during the procedure
  The airway pressure will be measured at the Y-piece by means of a differential pressure transducer
Pre-inspiratory potential at Electroencephalogram (EEG) | in real time, during the procedure
  Electroencephalogram (EEG) will be recorded using 30 surface electrodes (EEG international 10-20 system) (Rektor, 2002). Surface electrodes associated with ear lobes will serve as reference.
Arterial blood gas | in real time, during the procedure
  For patients with an arterial catheter, a blood gas analysis will be performed using an arterial blood sample of a volume of less than 1ml.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Pneumologie et Réanimation Médicale, Groupe Hospitalier Pitié Salpêtrière Paris, France, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lansing RW, Gracely RH, Banzett RB. The multiple dimensions of dyspnea: review and hypotheses. Respir Physiol Neurobiol. 2009 May 30;167(1):53-60. doi: 10.1016/j.resp.2008.07.012. Epub 2008 Jul 25. PMID 18706531
- [Result] Cherniack NS, Altose MD. Mechanisms of dyspnea. Clin Chest Med. 1987 Jun;8(2):207-14. PMID 3304811
- [Result] Morelot-Panzini C, Demoule A, Straus C, Zelter M, Derenne JP, Willer JC, Similowski T. Dyspnea as a noxious sensation: inspiratory threshold loading may trigger diffuse noxious inhibitory controls in humans. J Neurophysiol. 2007 Feb;97(2):1396-404. doi: 10.1152/jn.00116.2006. Epub 2006 Jul 26. PMID 16870842
- [Result] HAMMOND EC. SOME PRELIMINARY FINDINGS ON PHYSICAL COMPLAINTS FROM A PROSPECTIVE STUDY OF 1,064,004 MEN AND WOMEN. Am J Public Health Nations Health. 1964 Jan;54(1):11-23. doi: 10.2105/ajph.54.1.11. No abstract available. PMID 14117648
- [Result] Kessler R, Partridge MR, Miravitlles M, Cazzola M, Vogelmeier C, Leynaud D, Ostinelli J. Symptom variability in patients with severe COPD: a pan-European cross-sectional study. Eur Respir J. 2011 Feb;37(2):264-72. doi: 10.1183/09031936.00051110. Epub 2010 Nov 29. PMID 21115606
- [Result] Rabe KF, Hurd S, Anzueto A, Barnes PJ, Buist SA, Calverley P, Fukuchi Y, Jenkins C, Rodriguez-Roisin R, van Weel C, Zielinski J; Global Initiative for Chronic Obstructive Lung Disease. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2007 Sep 15;176(6):532-55. doi: 10.1164/rccm.200703-456SO. Epub 2007 May 16. PMID 17507545
- [Result] Nishimura K, Izumi T, Tsukino M, Oga T. Dyspnea is a better predictor of 5-year survival than airway obstruction in patients with COPD. Chest. 2002 May;121(5):1434-40. doi: 10.1378/chest.121.5.1434. PMID 12006425
- [Result] Celli BR, Cote CG, Marin JM, Casanova C, Montes de Oca M, Mendez RA, Pinto Plata V, Cabral HJ. The body-mass index, airflow obstruction, dyspnea, and exercise capacity index in chronic obstructive pulmonary disease. N Engl J Med. 2004 Mar 4;350(10):1005-12. doi: 10.1056/NEJMoa021322. PMID 14999112
- [Result] Esteban C, Quintana JM, Aburto M, Moraza J, Egurrola M, Perez-Izquierdo J, Aizpiri S, Aguirre U, Capelastegui A. Impact of changes in physical activity on health-related quality of life among patients with COPD. Eur Respir J. 2010 Aug;36(2):292-300. doi: 10.1183/09031936.00021409. Epub 2010 Jan 14. PMID 20075059
- [Result] Schmidt M, Demoule A, Polito A, Porchet R, Aboab J, Siami S, Morelot-Panzini C, Similowski T, Sharshar T. Dyspnea in mechanically ventilated critically ill patients. Crit Care Med. 2011 Sep;39(9):2059-65. doi: 10.1097/CCM.0b013e31821e8779. PMID 21572329
- [Result] Wilson PR. Clinical practice guideline: acute pain management. Clin J Pain. 1992 Sep;8(3):187-8. doi: 10.1097/00002508-199209000-00001. No abstract available. PMID 1421731
- [Result] Pochard F, Lanore JJ, Bellivier F, Ferrand I, Mira JP, Belghith M, Brunet F, Dhainaut JF. Subjective psychological status of severely ill patients discharged from mechanical ventilation. Clin Intensive Care. 1995;6(2):57-61. PMID 10150800
- [Result] de Miranda S, Pochard F, Chaize M, Megarbane B, Cuvelier A, Bele N, Gonzalez-Bermejo J, Aboab J, Lautrette A, Lemiale V, Roche N, Thirion M, Chevret S, Schlemmer B, Similowski T, Azoulay E. Postintensive care unit psychological burden in patients with chronic obstructive pulmonary disease and informal caregivers: A multicenter study. Crit Care Med. 2011 Jan;39(1):112-8. doi: 10.1097/CCM.0b013e3181feb824. PMID 21037472
- [Result] Pennock BE, Crawshaw L, Maher T, Price T, Kaplan PD. Distressful events in the ICU as perceived by patients recovering from coronary artery bypass surgery. Heart Lung. 1994 Jul-Aug;23(4):323-7. PMID 7960858
- [Result] van de Leur JP, van der Schans CP, Loef BG, Deelman BG, Geertzen JH, Zwaveling JH. Discomfort and factual recollection in intensive care unit patients. Crit Care. 2004 Dec;8(6):R467-73. doi: 10.1186/cc2976. Epub 2004 Oct 28. PMID 15566593
- [Result] Rotondi AJ, Chelluri L, Sirio C, Mendelsohn A, Schulz R, Belle S, Im K, Donahoe M, Pinsky MR. Patients' recollections of stressful experiences while receiving prolonged mechanical ventilation in an intensive care unit. Crit Care Med. 2002 Apr;30(4):746-52. doi: 10.1097/00003246-200204000-00004. PMID 11940739
- [Result] Cuthbertson BH, Hull A, Strachan M, Scott J. Post-traumatic stress disorder after critical illness requiring general intensive care. Intensive Care Med. 2004 Mar;30(3):450-5. doi: 10.1007/s00134-003-2004-8. Epub 2003 Sep 5. PMID 12961065
- [Result] Campbell ML, Templin T, Walch J. A Respiratory Distress Observation Scale for patients unable to self-report dyspnea. J Palliat Med. 2010 Mar;13(3):285-90. doi: 10.1089/jpm.2009.0229. PMID 20078243
- [Result] Campbell ML. Respiratory distress: a model of responses and behaviors to an asphyxial threat for patients who are unable to self-report. Heart Lung. 2008 Jan-Feb;37(1):54-60. doi: 10.1016/j.hrtlng.2007.05.007. PMID 18206527
- [Result] Persichini R, Gay F, Schmidt M, Mayaux J, Demoule A, Morelot-Panzini C, Similowski T. Diagnostic Accuracy of Respiratory Distress Observation Scales as Surrogates of Dyspnea Self-report in Intensive Care Unit Patients. Anesthesiology. 2015 Oct;123(4):830-7. doi: 10.1097/ALN.0000000000000805. PMID 26259140
- [Result] Hug F, Raux M, Morelot-Panzini C, Similowski T. Surface EMG to assess and quantify upper airway dilators activity during non-invasive ventilation. Respir Physiol Neurobiol. 2011 Sep 15;178(2):341-5. doi: 10.1016/j.resp.2011.06.007. Epub 2011 Jun 15. PMID 21699998
- [Result] Ward ME, Corbeil C, Gibbons W, Newman S, Macklem PT. Optimization of respiratory muscle relaxation during mechanical ventilation. Anesthesiology. 1988 Jul;69(1):29-35. doi: 10.1097/00000542-198807000-00005. PMID 3389564
- [Result] Parthasarathy S, Jubran A, Laghi F, Tobin MJ. Sternomastoid, rib cage, and expiratory muscle activity during weaning failure. J Appl Physiol (1985). 2007 Jul;103(1):140-7. doi: 10.1152/japplphysiol.00904.2006. Epub 2007 Mar 29. PMID 17395760
- [Result] Schmidt M, Chiti L, Hug F, Demoule A, Similowski T. Surface electromyogram of inspiratory muscles: a possible routine monitoring tool in the intensive care unit. Br J Anaesth. 2011 Jun;106(6):913-4. doi: 10.1093/bja/aer141. No abstract available. PMID 21576107
- [Result] Schmidt M, Kindler F, Gottfried SB, Raux M, Hug F, Similowski T, Demoule A. Dyspnea and surface inspiratory electromyograms in mechanically ventilated patients. Intensive Care Med. 2013 Aug;39(8):1368-76. doi: 10.1007/s00134-013-2910-3. Epub 2013 Apr 11. PMID 23575612
- [Result] Raux M, Straus C, Redolfi S, Morelot-Panzini C, Couturier A, Hug F, Similowski T. Electroencephalographic evidence for pre-motor cortex activation during inspiratory loading in humans. J Physiol. 2007 Jan 15;578(Pt 2):569-78. doi: 10.1113/jphysiol.2006.120246. Epub 2006 Nov 16. PMID 17110415
- [Result] Raux M, Ray P, Prella M, Duguet A, Demoule A, Similowski T. Cerebral cortex activation during experimentally induced ventilator fighting in normal humans receiving noninvasive mechanical ventilation. Anesthesiology. 2007 Nov;107(5):746-55. doi: 10.1097/01.anes.0000287005.58761.e8. PMID 18073550
- [Derived] Decavele M, Bureau C, Campion S, Nierat MC, Rivals I, Wattiez N, Faure M, Mayaux J, Morawiec E, Raux M, Similowski T, Demoule A. Interventions Relieving Dyspnea in Intubated Patients Show Responsiveness of the Mechanical Ventilation-Respiratory Distress Observation Scale. Am J Respir Crit Care Med. 2023 Jul 1;208(1):39-48. doi: 10.1164/rccm.202301-0188OC. PMID 36973007